CLINICAL TRIAL: NCT05172986
Title: Enhanced Recovery Program After a Robotic-assisted Surgery (RAAC) of Radical Prostatectomy. PROSTA-RAAC
Acronym: PROSTA-RAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A03292-37
Record Dates: First submitted 2021-12-21; First posted 2021-12-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer; Quality of Life; Recovery Programm
Keywords: Robotic assisted
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAAC (Program Arm) (Experimental): Patient under RAAC Program
  Interventions: Behavioral: Follow-up patient program
- Standard Arm (No Intervention): Standard patient procedure

INTERVENTIONS:
Behavioral: Follow-up patient program — An additional paramedical visit will be carried out before the surgery. The interview is carried out by the healthcare team. An organization within the service has been set up so that a nurse can be totally seconded for the RAAC mission. The consultation lasts 30 to 45 minutes.
  Arms: RAAC (Program Arm)

SUMMARY:
There are few published data on the benefit of Enhanced recovery program in radical prostatectomy in the management of localized prostate cancer. All the studies available on the subject are retrospective (1-3).

This randomized comparative study is proposed in order to compare in a homogeneous population (place and time) the interest of RAAC specifically in this surgery.

DETAILED DESCRIPTION:
The implementation of RAAC programs in healthcare establishments would improve the quality and safety of patient care (functional development and rapid convalescence of patients and reduction in postoperative morbidity through active prevention of perioperative complications) and optimization of care costs for health establishments and for health insurance (reduction in length of stay and convalescence, reduction in postoperative complications). Its implementation requires a strong involvement of all the teams and a transversal and multidisciplinary coordination, specifically dedicated to one type of intervention. This approach must therefore show its effectiveness by specialty and then by pathology within the same specialty.

There are few published data on the benefit of RAAC in radical prostatectomy in the management of localized prostate cancer. All the studies available on the subject are retrospective (1-3).

This randomized comparative study is proposed in order to compare in a homogeneous population (place and time) the interest of RAAC specifically in this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male over 40 and under 75
* Patient scheduled for a robot assisted radical prostatectomy within the center
* Affiliation to a social security scheme or beneficiary of such a scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Minor, age ≤ 40 years or ≥ 75 years
* ASA 4 or more
* Severe or poorly balanced associated conditions
* Covid + declared in the previous 3 months
* Refusal to participate in the study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative stay of RAAC-type treatment | 5 days
  To assess the length of postoperative stay of RAAC-type treatment compared to standard treatment, during a robotic-assisted radical prostatectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Augustin, Bordeaux, Nouvelle-Aquitaine, France

REFERENCES:
- [Derived] Pierquet G, Prevost E, Lopez L, Gaston R, Rouffilange J, Riviere J, Roche JB, Vuong N, Genty A, Hoepffner JL, Asimakopoulos AD, Piechaud PT. Enhanced recovery after surgery protocol does not reduce the length of postoperative hospitalization after robot-assisted radical prostatectomy. Outcomes from the first randomized controlled trial: the (PROSTA-RAAC) study. World J Urol. 2025 Nov 15;43(1):699. doi: 10.1007/s00345-025-06078-2. PMID 41240114